CLINICAL TRIAL: NCT02769117
Title: Utilizing Bone Ultrasound to Access Fracture Healing
Brief Title: Bone Ultrasound to Access Fracture Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Todd A. Milbrandt, M.D., Associate Professor of Orthopedics and Pediatrics,, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-008523
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Forearm Fracture; Clavicle Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound on fractured bone (Active Comparator): An ultrasound technique will be used to record the acoustic response of the fractured bone at each clinical visit until the fracture is healed. The ultrasound probe and a small hydrophone are placed on the exposed portion of the forearm on either sides of the fracture. The ultrasound intensity will be at the safe level according to the FDA regulation. Investigators will conduct the tests on the fracture and on the unaffected (contralateral) bone as the control. Typically this is at 1-, 2-, 4-, and 6- weeks following the fracture.
  Interventions: Procedure: Ultrasound on fractured bone
- Ultrasound on contralateral intact bone (Active Comparator): An ultrasound technique will be used to record the acoustic response of the intact bone as control at each clinical visit. The ultrasound probe and a small hydrophone are placed on the exposed portion of the forearm or clavicle. The ultrasound intensity will be at the safe level according to the FDA regulation. Investigators will conduct the tests on the fractured forearm/clavicle and on the unaffected (contralateral) forearm/clavicle as the control. Typically this is at 1-, 2-, 4-, and 6- weeks following the fracture.
  Interventions: Procedure: Ultrasound on contralateral intact bone

INTERVENTIONS:
Procedure: Ultrasound on fractured bone — A new ultrasound technique for children and adults who have sustained forearm or clavicle fractures
  Arms: Ultrasound on fractured bone
Procedure: Ultrasound on contralateral intact bone — A new ultrasound technique for the intact bone as the control for children and adults who have sustained forearm or clavicle fractures
  Arms: Ultrasound on contralateral intact bone

SUMMARY:
The purpose of this study is to evaluate sequential fracture healing with radius/ulna fractures or clavicle fractures and compare ultrasound to radiographs.

DETAILED DESCRIPTION:
Investigators will recruit 60 pediatric and adult patients with complete radius, ulna and/or clavicle fractures and obtain ultrasound data from the fractured bones and the contralateral intact bone (as control) at each clinical visit. Ultrasound will be compared to radiographs. Completion of this aim will validate the concept and correlate clinical healing with ultrasound findings. For the ultrasound method, investigators will use ultrasound energy to produce a secondary mechanical vibration in bone that can be used to characterize the integrity of the bone. (This is in contrast with conventional sonography where ultrasound echoes are used to image the tissue.) The proposed method is based on the use of Ultrasound Radiation Force (URF) to excite the bone. URF is a "pushing" force exerted by ultrasound on an object. This force can be static, transient (pulse), or harmonic. Harmonic URF can be generated by modulating the amplitude of the ultrasound beam at a desired frequency. This force initiates bone vibration, where the frequency and amplitude of such vibrations depend on bone geometry and elastic properties. Hence, any fracture (or fracture repair) will alter the vibration pattern, thus enabling us to monitor fracture and fracture healing by analyzing such patterns.

ELIGIBILITY:
Inclusion Criteria:

* Forearm fractures and no patients with hemiplegia -OR-
* Clavicle fractures

Exclusion Criteria:

* Non-English speakers
* Known pregnancy

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-05; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Sequential fracture healing | 5 years
  Ultrasound results will be compared between the fractured and unaffected extremity. This comparison allows investigators to compensate for variations in bone size, geometry, and surrounding muscles, thus calibrating the measurements to individual patient. The hypothesis is that the acoustic response of the fractured bone approaches to that of the unaffected bone as the fracture heals. Therefore, by comparing the test results obtained from the fractured and unaffected bone it is possible to evaluate the status of bone fracture and its healing level. In this process, investigators will correlate the results of ultrasound tests to clinical findings (e.g., radiographs) to validate the results from the ultrasound tests.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Milbrandt, M.D., Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials